CLINICAL TRIAL: NCT06806748
Title: Observational Study of Recovery of Gait in Sub-acute Hemiplegic Stroke Patients
Brief Title: Gait Recovery After Stroke
Acronym: GRAS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Strathclyde (Other)
Responsible Party: Sponsor
Other Study IDs: UoS_GRAS_2025
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Observational, gait, symmetry
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this observational study is to track the recovery of stance duration symmetry during the first 6 months after stroke using wearable sensors and explore the influence of stroke specific factors (time since stroke, stroke type, location and paretic side).

DETAILED DESCRIPTION:
Gait impairments can limit the ability to perform daily activities and increase the risk of falls in stroke survivors. Although rehabilitation improves walking in people with stroke, it is unclear whether the improvement relies on compensatory strategies or can be further improved to achieve normal or closer to normal performance.

Stance duration symmetry is an ideal measure of gait recovery in stroke survivors as it indicates the paretic sides capacity to control body weight and maintain balance during walking. Measuring stance duration symmetry may, therefore, be useful for monitoring gait recovery and could be considered as one of key goals in stroke rehabilitation.

Understanding the mechanisms of gait recovery in people with stroke is, therefore, essential for designing treatment program, setting realistic goals and appropriate timing for promoted intervention according to their stroke characteristics.

Our plan is to track changes in the symmetry of stance duration of hemiplegic patients during the first 6 months after stroke attached at the following time points: 1) at recruitment (within 2 weeks after of stroke), 2) 4th weeks (1 month) after stroke, 3) 12th weeks (3 months) after stroke, and 4) 26th weeks (6 months) after stroke. Two wearable accelerometers (the ActivPAL4+, PAL technology, Glasgow, UK) directly to the skin of both anterior thighs using sticky pads for 4 days (24 hours) period. Demographic (age and gender) and relevant clinical data (10-meter walk test, Modified Rivermead Mobility Index (RMI), stroke type, paretic side) will also be recorded as factors to explain gait symmetry.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* diagnosis of a first occurrence of stroke by consultant stroke physician
* Medically stable
* referred for rehabilitation
* functional ambulatory category of 1 and over

Exclusion Criteria:

* acute skin condition
* transient ischemic stroke
* comorbidities that may interfere with walking function, such as Parkinson's disease or lower limb amputation
* severe communication impairments or delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sub-acute stroke patients with hemiplegia who are referred for rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Gait symmetry | From enrollment to 6 months
  Gait symmetry will be measured from the signals produced by two thigh mounted inertial motion units. The variable of prime interest is the difference in stance duration between the hemiplegic and non-hemiplegic sides

SECONDARY OUTCOMES:
Rivermead Mobility Index | From enrollment to 6 months
  Standard, patient reported outcome measure of mobility
Ten meter walk test | From enrollment to 6 months
  Time it takes to walk 10 m. This is a well used, standardized objective test of mobility

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kerr, Ph.D, Principal Investigator — University of Strathclyde